CLINICAL TRIAL: NCT03147612
Title: Phase II Study of the Sequential Combination of Low-Intensity Chemotherapy and Ponatinib Followed by Blinatumomab and Ponatinib in Patients With Philadelphia Chromosome (Ph)-Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Low-Intensity Chemotherapy, Ponatinib and Blinatumomab in Treating Patients With Philadelphia Chromosome-Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0402; NCI-2018-01186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0402 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia With BCR-ABL1; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cyclophosphamide; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Methotrexate; merphos; pegfilgrastim; ponatinib; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, ponatinib, blinatumomab) (Experimental): See Detailed Description.
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Biological: Filgrastim; Drug: Methotrexate; Biological: Pegfilgrastim; Drug: Ponatinib; Biological: Rituximab; Drug: Vincristine

INTERVENTIONS:
Biological: Blinatumomab — Given via central catheter
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given intrathecally or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: Filgrastim-aafi; G-CSF; Neupogen; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Methotrexate — Given intrathecally or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial studies how well low-intensity chemotherapy and ponatinib work in treating patients with Philadelphia chromosome-positive and/or BCR-ABL positive acute lymphoblastic leukemia that may have come back or is not responding to treatment. Drugs used in chemotherapy, such as cyclophosphamide, vincristine, dexamethasone, methotrexate, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with rituximab and blinatumomab, may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Ponatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Granulocyte colony stimulating factor helps the bone marrow make recover after treatment. Giving low-intensity chemotherapy, ponatinib, and blinatumomab may work better in treating patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete molecular response (CMR) rate of ponatinib and blinatumomab in combination with low-intensity chemotherapy in patients with newly diagnosed Philadelphia chromosome (Ph)-positive and/or BAR-ABL-positive acute lymphoblastic leukemia (ALL). (Cohort 1) II. To evaluate the overall response (OR; complete response [CR] + complete response with hematologic improvement [CRi]) in patients with relapsed/refractory disease. (Cohort 2)

SECONDARY OBJECTIVES:

I. To evaluate other clinical efficacy endpoints (complete cytogenetic response, complete molecular response [CMR] [for relapsed/refractory population], event-free survival and overall survival) and safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To characterize the role of ABL1 kinase domain mutations on treatment failure and relapse in patients with Ph+ ALL treated with hyper-CVD plus ponatinib and blinatumomab.

II. To determine the impact of recurrent genomic alterations and ribonucleic acid (RNA) expression at diagnosis on relapse free survival (RFS) in patients with Ph+ ALL treated with hyper-CVD plus ponatinib and blinatumomab.

III. To investigate the impact of next-generation sequencing-based minimal residual disease assessment on relapse-free survival in patients with Ph+ ALL.

IV. To determine the effect on immune cell subsets in patients with Ph+ ALL treated with blinatumomab plus ponatinib.

OUTLINE:

CYCLES 1 and 3: Patients receive ponatinib orally (PO) once daily (QD) on days 1-21 of cycle 1 and on days 1-28 of subsequent cycles, cyclophosphamide intravenously (IV) twice daily (BID) over 3 hours on days 1-3, rituximab IV over 4-6 hours on days 1 and 11, vincristine IV over 15 minutes on days 1 and 11, and pegfilgrastim or filgrastim subcutaneously (SC) daily on day 4. Patients also receive methotrexate intrathecally via spinal tap on day 2 and cytarabine intrathecally on day 7 in the absence of disease progression or unacceptable toxicity.

CYCLES 2 and 4: Patients receive ponatinib PO QD on days 1-28, methotrexate IV over 24 hours on day 1 and intrathecally on day 8, cytarabine IV BID over 2-3 hours on days 2 and 3 and intrathecally on day 5, pegfilgrastim or filgrastim SC daily on day 4, and rituximab IV over 4-6 hours on days 1 and 8 in the absence of disease progression or unacceptable toxicity.

CYCLES 5-8: Patients receive blinatumomab via central catheter continuously over weeks 1-4 every 6 weeks. Patients also receive methotrexate intrathecally on day 1 of cycle 5 and on day 8 of cycle 6 and cytarabine intrathecally on day 7 of cycle 5 and on day 1 of cycle 6 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY:

CYCLES 1-3, 5-7, 9-11, and 13-15: After 4 cycles of blinatumomab, if disease has not gotten worse, patients receive vincristine IV over 15 minutes on day 1, prednisone PO on days 1-5, and ponatinib PO QD on days 1-28.

CYCLES 4, 8, and 12: Patients receive blinatumomab via central catheter continuously over weeks 1-4 every 6 weeks and ponatinib PO QD on days 1-28.

Treatment repeats every 28 days for up to 15 cycles in the absence of disease progression or unacceptable toxicity. Patients unable to receive blinatumomab, you may receive maintenance therapy with vincristine, prednisone, and ponatinib for a total of about 24 cycles at the discretion of doctor.

POST-MAINTENANCE THERAPY: Patients receive ponatinib PO QD on days 1-28. Cycles repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age with previously untreated Ph-positive ALL (either t(9;22) and/or BCR-ABL positive) (includes patients initiated on first cycle of hyper-CVAD before cytogenetics known. These patients could have received one or two cycles of chemotherapy with or without other TKIs and still eligible.

  * If they achieved CR, they are assessable only for event-free and overall survival, or
  * If they failed to achieve CR, they are assessable for CR, event-free, and overall survival.

Patients >= 18 years of age with relapsed/refractory Ph-positive ALL or lymphoid accelerated or blast phase chronic myelogenous leukemia (CML)

* Performance status =< 2 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome
* Alanine aminotransferase (ALT) =< 3 x ULN
* Aspartate aminotransferase (AST) =< 3 x ULN
* Serum lipase and amylase =< 1.5 x ULN
* Creatinine =< 2.0 mg/dl
* Female patients who: are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who: agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Adequate cardiac function as assessed clinically by history and physical examination
* Signed informed consent

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Known active hepatitis B. Patients with chronic hepatitis B who are on appropriate viral suppressive therapy may be allowed after discussion with the principal investigator (PI)
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
* History of alcohol abuse
* Uncontrolled hypertriglyceridemia
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Uncontrolled, or active cardiovascular disease, specifically including, but not restricted to: myocardial infarction (MI), stroke, or revascularization within 3 months; unstable angina or transient ischemic attack; congestive heart failure prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment; diagnosed or suspected congenital long QT syndrome; clinically significant atrial or ventricular arrhythmias as determined by the treating physician; prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 470 msec) unless corrected after electrolyte replacement. or approved by cardiologist; Significant venous or arterial thromboembolism including deep venous thrombosis or pulmonary embolism. Patients with a history of treated prior superficial or catheter associated phlebitis will not be considered as significant embolism and after discussion with principal investigator (PI) will not be excluded from eligibility. Uncontrolled hypertension (diastolic blood pressure > 90 mmHg; systolic > 140mmHg). Patients with hypertension should be under treatment on study entry to effect blood pressure control
* Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days or 5 half-lives before the first dose of ponatinib in patients with newly diagnosed only
* History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. Patients with active CNS leukemia will NOT be excluded
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control
* History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); and diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients with documented significant pleural or pericardial effusions unless they are thought to be secondary to their leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Complete molecular response (CMR) in newly diagnosed Philadelphia chromosome (Ph)-positive and/or BCR-ABL-positive participants | Up to 84 days (3 courses)
  The CMR rate within the first 3 courses for cohort 1 or rate within the first 2 courses for cohort 2 will be estimated along with the 95% credible intervals. Similar analyses will be performed for estimating the rate of complete cytogenetic response and major molecular response rates.
Overall response (OR) in participants with relapsed/refractory acute lymphoblastic leukemia | Up to 6 years
  Overall response is defined as complete response (CR) + complete response with hematologic improvement (CRi) in participants with relapsed/refractory disease.

SECONDARY OUTCOMES:
Complete cytogenetic response | Up to 6 years
  Will be estimated along with the 95% credible intervals.
CMR for relapsed/refractory population | Up to 6 years
  Will be estimated along with the 95% credible intervals.
Event-free survival (EFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 6 years
  The Kaplan-Meier method will be used to assess EFS probabilities for each cohort.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up to 6 years
  The Kaplan-Meier method will be used to assess OS probabilities for each cohort.
Incidence of adverse events (AEs) | Up to 6 years
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org